CLINICAL TRIAL: NCT01175291
Title: Randomized, Double Blind Phase II Study of FOLFOX/Bevacizumab Combined With MK-0646 Versus FOLFOX/Bevacizumab Combined With Placebo in First-Line Treatment of Metastatic Colorectal Cancer
Brief Title: FOLFOX/Bevacizumab +/- MK-0646 in Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: treatment deemed ineffective so accrual was closed
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCC-16145
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colon; rectum; colorectal; metastatic; adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — dalotuzumab; Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - FOLFOX 7 + MK-0646 (Active Comparator)
  Interventions: Drug: MK-0646
- Arm B - FOLFOX 7 + Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-0646 — ARM A will receive FOLFOX 7 (Oxaliplatin with leucovorin + 5-Fluorouracil [5-FU] + Bevacizumab) + MK-0646 (Investigational).
  Other Names: oxaliplatin; leucovorin; 5-FU; Fluorouracil; bevacizumab
  Arms: Arm A - FOLFOX 7 + MK-0646
Drug: Placebo — ARM B will receive FOLFOX 7 (Oxaliplatin with leucovorin + 5-Fluorouracil [5-FU] + Bevacizumab) + placebo: standard of care chemotherapy plus placebo.
  Other Names: oxaliplatin; leucovorin; 5-FU; 5-Fluorouracil; bevacizumab
  Arms: Arm B - FOLFOX 7 + Placebo

SUMMARY:
The purpose is to study the efficacy (effectiveness) of a new drug, MK-0646, in metastatic colorectal cancer. MK-0646 is an investigational or experimental anti-cancer agent that has not yet been approved by the U.S. Food and Drug Administration (FDA) for use in metastatic colorectal cancer or any other disease.

This study will assess whether adding MK-0646 to an FDA-approved standard of care chemotherapy improves participants' duration of progression-free survival. MK-0646 is believed to inhibit the receptor of a protein called IGF-1 (Insulin-like Growth Factor) which is thought to contribute to cancer development and growth. However, there is no guarantee that MK-0646 will slow cancer development and growth.

Other purposes of this study include:

* looking at the safety and tolerability of MK-0646
* comparing MK-0646 + standard of care chemotherapy with placebo + standard of care chemotherapy (placebo is a substance that looks like an active drug but has no active ingredient) The standard of care chemotherapy in this study is called FOLFOX 7. FOLFOX 7 includes the drugs oxaliplatin with leucovorin, 5-Fluorouracil (5-FU), and bevacizumab.

DETAILED DESCRIPTION:
Participants randomized to ARM A will receive modified FOLFOX 7 every other week + MK-0646 every week:

5-FU 400 mg/m2 by intravenous infusion over 2-5 minutes Leucovorin 400 mg/m2 by intravenous infusion over 2 hours Oxaliplatin 85 mg/m2 by intravenous infusion over 2 hours (with leucovorin) Bevacizumab 5 mg/kg by intravenous infusion over 30 minutes (+/- 15 minutes) following infusions may be given over 10 minutes (+/- 10 minutes) if the first infusion is tolerated well.

5-FU 2400 mg/m2 by continuous intravenous infusion over 46 hours (may be delivered via automated outpatient pump) Antiemetics (drugs that prevent nausea and vomiting): 5-HT3 receptor antagonist (e.g. ondansetron) and dexamethasone are recommended prior to chemotherapy.

MK-0646 10 mg/kg by intravenous infusion over 60 minutes every week (participants larger than 100 kg [220 pounds] will receive their infusions over 120 minutes).

Participants randomized to ARM B will receive modified FOLFOX 7 every other week + placebo every week:

5-FU 400 mg/m2 by intravenous infusion over 2-5 minutes Leucovorin 400 mg/m2 by intravenous infusion over 2 hours Oxaliplatin 85 mg/m2 by intravenous infusion over 2 hours (with leucovorin) Bevacizumab 5 mg/kg by intravenous infusion over 30 minutes (+/- 15 minutes); following infusions may be given over 10 minutes (+/- 10 minutes) if the first infusion is tolerated well.

5-FU 2400 mg/m2 by continuous intravenous infusion over 46 hours (may be delivered via automated outpatient pump) Antiemetics: 5-HT3 receptor antagonist (e.g. ondansetron) and dexamethasone are recommended prior to chemotherapy Placebo by intravenous infusion over 60 minutes every week (participants larger than 100 kg [220 pounds] will receive their infusions over 120 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal adenocarcinoma.
* Measurable disease by RECIST criteria.
* Adequate hepatic function: total bilirubin ≤2.0 x upper limits of normal (ULN); Aspartate Amino Transferase (AST)/Alanine Amino Transferase (ALT) ≤3.0X upper limits of normal (or ≤5X upper limits of normal if attributable to liver metastases).
* Adequate renal function: serum creatinine ≤2.0 mg/dl.
* Adequate bone marrow function: absolute neutrophil count ≥1,500/mm3; platelets ≥ 100,000/mm3.
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) levels ≤1.5 upper limit of normal (unless patients receiving coumadin anticoagulation in which case a stable international normalized ratio (INR) of 2-3 is required).
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Life expectancy ≥ 12 weeks.
* Negative pregnancy test.
* Ability to sign informed consent.

Exclusion Criteria:

* Prior systemic chemotherapy for metastatic colorectal cancer
* Prior oxaliplatin in the adjuvant setting within 12 months
* Uncontrolled central nervous system metastases or carcinomatous meningitis.
* Myocardial infarction in the past 6 months.
* Major surgery within 8 weeks prior to enrollment.
* Uncontrolled serious medical or psychiatric illness.
* Inadequately controlled hypertension (defined as systolic blood pressure >160mmHg, or diastolic blood pressure > 100mmHg).
* Pregnant or lactating women. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of study.
* Prior experimental therapy targeting the IGF-1 pathway
* Concurrent malignancy (with the exception of squamous or basal cell skin carcinoma)
* Planned surgical metastasectomy
* Patient has known hypersensitivity to components of treatment, their analogs, or drugs of similar chemical or biologic composition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Average of 12 months
  To determine whether the administration of MK-0646 with FOLFOX and bevacizumab (experimental arm) improves progression-free survival (PFS) versus FOLFOX and bevacizumab combined with placebo (control arm).

SECONDARY OUTCOMES:
Objective Radiographic Response | Average of 12 months
  To determine whether the objective radiographic response (ORR) is higher in patients treated with FOLFOX and bevacizumab combined with MK-0646 (experimental arm) versus FOLFOX and bevacizumab combined with placebo (control arm).
Overall Survival | Average of 12 Months
  To determine whether overall survival (OS) is higher in patients treated with FOLFOX and bevacizumab combined with MK-0646 (experimental arm) versus FOLFOX and bevacizumab combined with placebo (control arm).
Number of Participants with Adverse Events | Average of 12 months
  To determine the safety and tolerability of MK-0646 combined with FOLFOX and bevacizumab. Safety and tolerability will be assessed according to the NIH/NCI CTC Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.